CLINICAL TRIAL: NCT06297811
Title: Efficacy and Safety of Trilaciclib in Myeloprotection During Chemotherapy for Advanced/Recurrent Malignant Solid Tumors - A Phase II Study
Brief Title: Myeloprotection With Trilaciclib in Pan-cancer Population
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Rui-hua Xu, MD, PhD, President and Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SMA PT 001
Record Dates: First submitted 2024-01-29; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Non-Small Cell Lung Cancer; Breast Cancer; Endometrial Cancer; Cervical Cancer; Head And Neck Squamous Cell Carcinomas
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — trilaciclib; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Trilaciclib group (Experimental)
  Interventions: Drug: Trilaciclib Injection; Drug: Paclitaxel; Drug: Carboplatin
- Control group (Active Comparator)
  Interventions: Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Trilaciclib Injection — Experimental: trilaciclib group Intervention: Drug: Trilaciclib Injection [Cosela] 240 mg/m^2, intravenous drip over 30 min within 4 hours before chemotherapy administration on the same day
  Arms: Trilaciclib group
Drug: Paclitaxel — Drug: Paclitaxel 175 mg/m^2, intravenous drip over ≥ 3 hours , d1, Q3W, at least 6 cycles.
Drug: Carboplatin — area under curve(AUC) 5~6, intravenous drip over ≥ 1 hours, d1, Q3W, at least 6 cycles.

SUMMARY:
The goal of this open-label randomized controlled study is to assess the myeloprotective effect of trilaciclib in pan-cancer population. The main questions it aims to answer are:

* effect and safety of trilaciclib on myeloprotection in cancer patients receiving paclitaxel plus carboplatin chemotherapy
* does trilaciclib 's myeloprotective efficacy in patients receiving the same chemotherapy regimen correlate with tumor type

Participants will be randomized 2:1 to the treatment arm of trilaciclib in combination with a paclitaxel and carboplatin-based regimen and the control arm of a paclitaxel and carboplatin-based regimen for at least 6 cycles or until disease progression or intolerable toxicity. Patients in both groups could extend the chemotherapy cycle at the investigator 's discretion depending on the tumor type and in combination with anti-angiogenic/PD-X/anti-HER2 therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Eastern Cooperative Oncology Group (ECOG) performance score 0-1;
3. Histologically or cytologically confirmed advanced or recurrent solid malignant tumors, including:

   * Unresectable stage III/IV non-small cell lung cancer (NSCLC);
   * Recurrent or metastatic breast cancer (BC);
   * Newly diagnosed International Federation of Gynecology and Obstetrics (FIGO) stage IC-IV epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer without further surgical planning before disease progression; or recurrent platinum-sensitive ovarian cancer (OC);
   * FIGO stage III-IV or recurrent endometrial cancer (EC), including endometrioid carcinoma and serous or clear cell carcinoma;
   * FIGO stage IVB (including persistent) or recurrent cervical cancer (CC) (≤ 1 prior platinum-based therapy) not amenable to radical surgery or radiotherapy;
   * Recurrent or metastatic head and neck squamous cell carcinoma (HNSCC) (including primary lesions located in the larynx, oropharynx, hypopharynx, oral cavity, undifferentiated or poorly differentiated nasopharyngeal carcinoma, and salivary gland carcinoma), which is not suitable for further surgery or radiotherapy.
4. At least one measurable lesion according to RECIST version 1.1;
5. Received up to one prior systemic chemotherapy and no prior paclitaxel plus carboplatin chemotherapy;
6. Adequate organ function meeting the following criteria: (1) adequate bone marrow function: Hb ≥ 100 g/L (no ESA or blood transfusion within 14 days before the first dose); ANC ≥ 2 × 10^9/L (no G-CSF within 14 days before the first dose); platelet count ≥ 100 × 10^9/L (no rhTPO, rhIL-11 or platelet transfusion within 14 days before the first dose); (2) adequate liver and kidney function: alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN), aspartate aminotransferase (AST) ≤ 2.5 × ULN, total bilirubin (TBIL) ≤ 1.5 × ULN, serum creatinine ≤ 1.5 × ULN, endogenous creatinine clearance > 50 ml/min (Cockcroft-Gault formula); (3) adequate cardiac function: left ventricular ejection fraction (LVEF) ≥ 55%;
7. Life expectancy ≥ 3 months;
8. Females of childbearing potential agree to practice reliable contraception during the clinical trial and have a negative serum or urine pregnancy test within 7 days prior to dosing;
9. Voluntarily join this study, sign informed consent, have good compliance and are willing to cooperate with follow-up.

Exclusion Criteria:

1. History of myeloid leukemia, myelodysplastic syndrome, or concomitant sickle cell disease;
2. Symptomatic CNS metastases and/or leptomeningeal disease requiring immediate radiation or steroid therapy;
3. Received surgery or radiotherapy within 4 weeks prior to the first dose of study drug;
4. Receipt of any investigational drug ≤ 30 days or ≤ 5 half-lives (whichever is longer) prior to the first dose of study drug;
5. Platinum-resistant OC (refractory to 1 line of platinum-based chemotherapy or recurrent platinum-based chemotherapy within 6 months prior to the first dose of study drug);
6. Requires concurrent radiotherapy;
7. Known history of hypersensitivity to the drug components of this protocol;
8. Pregnant or lactating women;
9. Any other condition that, in the opinion of the investigator, would make the patient inappropriate for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of grade 3/4 neutropenia within 6 cycles | Up to 18 weeks
  Percentage of patients with at least one absolute neutrophil count (ANC) < 1.0 × 10 ^ 9/L in total number of patients included in the analysis set.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Oncology,Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China